CLINICAL TRIAL: NCT03355534
Title: Effect of Dexmedetomidine on Maintenance and Recovery of Cranial Aneurysm Surgery
Brief Title: Dexmedetomidine Improves Recovery After Cranial Aneurysm Surgery
Acronym: DACA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhihong LU (Other)
Responsible Party: Sponsor-Investigator, Zhihong LU, clinical professor, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: XJH-A-2017-10-10
Record Dates: First submitted 2017-11-19; First posted 2017-11-28 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Aneurysm Cerebral
Keywords: dexmedetomidine; general anesthesia; cerebral aneurysm
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- nasal dexmedetomidine (Experimental): dexmedetomidine is given nasally, saline is given intravenously
  Interventions: Drug: nasal dexmedetomidine; Drug: intravenous saline
- intravenous dexmedetomidine (Experimental): saline is given nasally, dexmedetomidine is given intravenously
  Interventions: Drug: Intravenous dexmedetomidine; Drug: nasal saline
- normal saline (Placebo Comparator): saline is given nasally and intravenously
  Interventions: Drug: intravenous saline; Drug: nasal saline

INTERVENTIONS:
Drug: Intravenous dexmedetomidine — drug is intravenously infused to patients
  Arms: intravenous dexmedetomidine
Drug: nasal dexmedetomidine — drug is nasally given to patients
  Arms: nasal dexmedetomidine
Drug: intravenous saline — saline is given to patients intravenously
  Arms: nasal dexmedetomidine; normal saline
Drug: nasal saline — normal saline is given to patients nasally
  Arms: intravenous dexmedetomidine; normal saline

SUMMARY:
Dexmedetomidine induces analgesic and sedative effects and is reported to decrease agitation during emergence after general anesthesia in various surgeries. For patients undergoing cranial aneurysm surgeries, a calm anesthesia and emergence is important. In this study, the investigatorstend to observe the effect of dexmedetomidine on maintenance and recovery of patients undergoing cranial aneurysm surgeries.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cerebral aneurysm embolism under general anesthesia

Exclusion Criteria:

* patients with bradycardia or atrioventricular heart block
* patients with ASA(American Society of Anesthesiologists) status over 3
* patients with body mass index(BMI)≥30kg/m2
* patients with difficulty in communication
* patients with ruptured aneurysm
* patients suspected or proved to be pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
incidence of coughing | from end of infusing anesthetics to 2 minutes after extubation, averagely 30 minutes

SECONDARY OUTCOMES:
Ricker's agitation-sedation score | from end of infusing anesthetics to 2 minutes after extubation, averagely 30 minutes
score of coughing | from end of infusing anesthetics to 2 minutes after extubation, averagely 30 minutes
  0=no coughing;1=intermittent coughing;2=continuous coughing
time to response to verbal command | from end of infusing anesthetics to response to verbal command,averagely 20 minutes
time to extubation | from end of infusing anesthetics to extubation,averagely 28 minutes
blood pressure before and after extubation | from end of infusing anesthetics to 2 minutes after extubation, averagely 30 minutes
blood glucose before and after aneurysm embolism | immediately before inserting coil and after finishing inserting coil,an average of 1 hour
blood lactate before and after aneurysm embolism | immediately before inserting coil and after finishing inserting coil,,an average of 1 hour
Mini-mental state examination score | 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lize Xiong, Study Chair — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Peng K, Wu S, Liu H, Ji F. Dexmedetomidine as an anesthetic adjuvant for intracranial procedures: meta-analysis of randomized controlled trials. J Clin Neurosci. 2014 Nov;21(11):1951-8. doi: 10.1016/j.jocn.2014.02.023. Epub 2014 Jun 25. PMID 24974190
- [Result] Soliman RN, Hassan AR, Rashwan AM, Omar AM. Prospective, randomized controlled study to assess the role of dexmedetomidine in patients with supratentorial tumors undergoing craniotomy under general anesthesia. Middle East J Anaesthesiol. 2011 Feb;21(1):23-33. PMID 21991729
- [Result] Elbakry AE, Ibrahim E. Propofol-dexmedetomidine versus propofol-remifentanil conscious sedation for awake craniotomy during epilepsy surgery. Minerva Anestesiol. 2017 Dec;83(12):1248-1254. doi: 10.23736/S0375-9393.17.11873-0. Epub 2017 Jun 14. PMID 28631453
- [Result] Jun JH, Kim KN, Kim JY, Song SM. The effects of intranasal dexmedetomidine premedication in children: a systematic review and meta-analysis. Can J Anaesth. 2017 Sep;64(9):947-961. doi: 10.1007/s12630-017-0917-x. Epub 2017 Jun 21. PMID 28639236
- [Result] Sun Y, Li Y, Sun Y, Wang X, Ye H, Yuan X. Dexmedetomidine Effect on Emergence Agitation and Delirium in Children Undergoing Laparoscopic Hernia Repair: a Preliminary Study. J Int Med Res. 2017 Jun;45(3):973-983. doi: 10.1177/0300060517699467. Epub 2017 Mar 21. PMID 28470100